CLINICAL TRIAL: NCT03983213
Title: The Clinical, Radiological, Isokinetic Assessment With Gait Analysis in Children After Surgical Treatment of Patellar Recurrent Dislocation.
Brief Title: The Comprehensive Assessment in Children After Surgical Treatment of Patellar Recurrent Dislocation.
Status: Completed | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-BCO.34/2019
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Patellar Dislocation; Patellar Instability
Keywords: Patellar instability; Recurrent patellar dislocation; Isokinetics; Children; MPFL reconstruction
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pat. after mpfl reconstruction: All 45 subjects operated with mpfl reconstruction included to chek-up after follow-up.
  Interventions: Procedure: mpfl reconstruction

INTERVENTIONS:
Procedure: mpfl reconstruction — Harvested gracilis tendon is pulled through patella and femur in anatomic position and locked with interference screw.

SUMMARY:
The aim of this prospective study is to assess extension apparatus function of the knee based on clinical, radiological, isokinetic and gait analysis data in patients after surgical treatment. There will be used physical examination, Lysholm-Tegner and Kujala scale for clinical assessment. Merchant and lateral X-ray pictures will be analysed for patellar position verification along with isokinetic and gait evaluation to produce conclusions referring to efficacy of the treatment. All subjects included in the study were treated with mpfl reconstruction. Follow-up longer than 2 years in all cases, about 45 patients included.

DETAILED DESCRIPTION:
Recurrent patellar dislocation occurs mostly in adolescents. Recently medial patellofemoral ligament reconstruction has become treatment of choice in most cases. There is still insufficient literature to assess the operative treatment results according to functional testing.

The aim of this prospective study is to assess extension apparatus function of the knee based on clinical, radiological, isokinetic and gait analysis data in patients after surgical treatment. There will be used physical examination, Lysholm-Tegner and Kujala scale for clinical assessment. Merchant and lateral X-ray pictures will be analysed for patellar position verification along with isokinetic and gait evaluation to produce conclusions referring to efficacy of the treatment. All subjects included in the study were treated with mpfl reconstruction with gracilis tendon harvesting. Follow-up provided is longer than 2 years in all 45 cases planned to enroll. All subject are to be mailed and invited to check-up visit including analysis of parameters mentioned above. Soon after data collection text of the publication will be made. The results will be discussed with recent literature and conclusions will be made.

ELIGIBILITY:
Inclusion Criteria:

* age <18 yo
* recurrent patellar dislocation
* ready for follow-up

Exclusion Criteria:

* age <18 yo
* osteochondral fracture
* habitual dislocation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 45 patients under 18 yo, 30 females, 15 males, average age of 15 yo
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Dislocation recurrence | 2 years
  The incident of patellar dislocation after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kryspin Niedzielski, Ph.D., Study Chair — Polish Mother Memorial Hospital Research Institute; Krzysztof Małecki, Ph.D., Study Director — Polish Mother Memorial Hospital Research Institute; Jacek Beczkowski, M.D., Principal Investigator — Polish Mother Memorial Hospital Research Institute; Paweł Flont, Ph. D., Principal Investigator — Polish Mother Memorial Hospital Research Institute
Locations (1):
- Polish Mother Memorial Hospital Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
Sharing IPD after data collection in Exel
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After data collection
Access Criteria: Not known yet